CLINICAL TRIAL: NCT06173687
Title: Feasibility, Prospective, Multicentric, Cross-sectional Investigation to Characterize Daily Impedance Fluctuations and Satisfaction in Challenging Listening Environments in Experienced Adult CI Recipients Using the Mobile Research App (MRA)
Brief Title: Multi-center Study to Examine Changes to the Environment Surrounding the Electrodes in the Cochlea and to Capture the Most Challenging Listening Environments Experienced by Persons With a Cochlear Implant
Acronym: DICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AI5846
Record Dates: First submitted 2023-10-19; First posted 2023-12-18 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental)
  Interventions: Device: The impedance measurement task using the Mobile Research App (MRA)

INTERVENTIONS:
Device: The impedance measurement task using the Mobile Research App (MRA) — Characterisation of impedance and real-world monitoring of hearing difficulty in range of listening environments.

SUMMARY:
This early feasibility study aims to collect pilot data on impedance measurements in real-world environments and to collect real-world and difficult listening situations and the factors impacting this, reflecting situations the subjects encounter during their daily life outside of the clinic. Improving the monitoring of both aspects may lead to improvements in monitoring and personalising the fitting to optimise hearing outcomes for persons with a cochlear implant.

DETAILED DESCRIPTION:
This is a feasibility, prospective, multi-country, multi-centre, cross-sectional interventional clinical investigation in adults with a CE labelled cochlear implant.

No Randomisation nor blinding to avoid bias is applicable in this study since there is no comparator.

Subjects will attend two scheduled study visits over a two-month study period. At and in between study visits, subjects will undergo hearing assessments and safety monitoring. The subjects will perform daily impedance test tasks and complete a questionnaire in order to obtain the first primary endpoint, i.e. characterization of Daily Impedance Fluctuations.

Furthermore, the subjects will do EMA tasks to obtain the secondary objectives to capture daily-life, real-world listening environments and challenging listening environments.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older (no upper age limit).
* Implanted with CIC4-based implant with a Contour Advance, Slim Straight or Slim Modiolar electrode array with at least 6 months experience.
* Candidate is a fluent speaker in the language used to assess speech perception performance, as determined by the investigator.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Score below 3 on the screening subset of questions from the Mobile Device Proficiency Questionnaire (digital literacy check).
* A failed ECE1 or ECE2 (i.e. flagged, open circuit or short circuit)
* Additional health factors, known to the investigator, that would prevent or restrict participation in the evaluations, including significant visual impairment and/or dexterity issues.
* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
* Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation.
* Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless the other investigation was/is a Cochlear sponsored investigation and determined by the investigator or Sponsor to not impact this investigation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (2):
  - Cochlear Macquarie, Sydney, New South Wales
  - HEARnet, Carlton, Victoria
- ENT Department, Sint-Augutinus Antwerp, Wilrijk, Antwerp, Belgium
- Cochlear Bone Anchored Solutions AB (CBAS), Mölnlycke, Västergötland, Sweden

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for public sharing of IPD collected in this study. Data may be provided to individual researchers on request.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 51
Completed | 45
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 51
Age, Continuous [Median (Full Range); unit: years] | 65 [28 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Cochlear implant experience [Median (Full Range); unit: years] | 5.7 [0.6 to 18.8]

OUTCOME MEASURES:

1. Primary Outcome: Impedance Measurements
Description: Median of the standard deviation in total electrode impedance (measured in kOhm, averaged across 22 electrode contacts) between days for 8 weeks.
Time Frame: 8 Weeks
Measure: Median (Inter-Quartile Range); unit: kOhm
Arm/Group | All Participants
Number analyzed (Participants) | 44
kOhm | 0.36 [0.27 to 0.67]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 3/51
Other Adverse Events (participants affected / at risk) | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=51)
Tachycardia (Cardiac disorders) | 1
Epileptic seizures (Nervous system disorders) | 1
Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT06173687/Prot_SAP_000.pdf